CLINICAL TRIAL: NCT01281241
Title: The Connection Between Mechanical Alternans Measured by Pressure-Volume (PV) Loop Catheter in Patients With Ischemic Heart Failure and the Occurrence of Microvolt T Wave Alternans (MTWA)
Brief Title: Study on Mechanical and Electrical Alternans
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: A.A.M Wilde, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Other Study IDs: NL33244.018.10
Record Dates: First submitted 2011-01-20; First posted 2011-01-21 (Estimated); Last update posted 2011-01-21 (Estimated); Status verified 2010-10

CONDITIONS: Heart Failure; Ischemia; Ventricular Arrhythmia
Keywords: MTWA; mechanical alternans
MeSH Terms: conditions — Heart Failure; Ischemia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The main objective is to investigate mechanical alternans and MTWA in patients with heart failure caused by coronary artery disease to demonstrate a possible correlation between these two phenomena.

DETAILED DESCRIPTION:
In patients with severe heart failure and aortic valve disease mechanical alternans or pulsus alternans (a condition in which there is a beat-to-beat oscillation in the strength of cardiac muscle at a constant heart rate) is observed.

The mechanisms linking mechanical to electrophysiological dysfunction in heart failure are still under investigation, but impaired calcium cycling is the most striking abnormality of failing myocytes, and is most responsible for contractile dysfunction. Yet it remains unclear how this influences susceptibility to arrhythmias.

The MTWA is suggested as a risk marker to identify high risk patients for potential VTEs but the underlying mechanism is not completely understood. The aim of this study is to investigate this in a clinical setting by measuring LV parameters using a PV loop conductance catheter and generate TWA recording simultaneously to demonstrate a possible correlation between these two phenomena in patients with ischemic heart failure and find out if MTWA could turn into a more valuable risk factor.

Our hypothesis is that alternating changes in LV filling explains the electrocardiogenesis of TWA by changing the position of the heart relative to the body surface electrodes in an alternating way.

ELIGIBILITY:
Inclusion Criteria:

* Patients with heart failure caused by coronary artery disease
* Indication for left ventricular radiofrequency (LV RF) ablation
* LVEF ≤ 35% measured by echocardiogram or MRI

Exclusion Criteria:

* hemodynamically instable patients
* age under 18 and over 85 years,
* heart failure not caused by coronary artery disease
* Severe co-morbidity

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to the hospital with a left ventricular ejection fraction (LVEF) under 35%, due to coronary artery disease with an indication for electrophysiological investigation.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2010-09; Primary Completion 2011-12 (Estimated); Study Completion 2012-06 (Estimated)

PRIMARY OUTCOMES:
Presence or absence of mechanical alternans and MTWA | 1 year

SECONDARY OUTCOMES:
Differences in reduced or more preserved LVEF and the occurrence of the two phenomena | 1 year
The occurrence of ventricular tachyarrhythmic events. | 1 year
Influence of LV compliance on arrhythmogenesis of the infarction border zone. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Arthur AM Wilde, MD, PhD, Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Locations (1):
- Academic Medical Center, Amsterdam, Netherlands